CLINICAL TRIAL: NCT04823078
Title: Effects of Activity Based Therapy on Upper Limb Strength and Transfer in Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/1009 Namra Urooj
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity base therapy (Active Comparator)
  Interventions: Other: Activity base therapy
- Strength training (Other)
  Interventions: Other: Strength training

INTERVENTIONS:
Other: Activity base therapy — activity based therapy
  Weight bearing activities of daily living like vertical lifting, bilateral body weight shifting, lifting and shifting, forward reaching and sideways reaching.
  Arms: Activity base therapy
Other: Strength training — Strengthening exercises of upper limb involved muscles (elbow extensors, shoulder adductors, abductors, wrist extensors, shoulder protractors and retractors
  Arms: Strength training

SUMMARY:
In our society spinal cord injury is a major problem.activity based therapy and conventional therapy has a potentional to improve upper limb strength and transfer in tetraplegic patients.

The aim of this study is to determine the effects of activity based therapy versus conventional therapy to improve the upper limb strength and transfer in spinal cord injury.

The study design used was randomized clinical trial. The study was conducted at the paraplegic center Peshawar in 6 weeks after the approval of synopsis. A sample size of 16 participants was taken with complete and incomplete spinal cord injury received using lottery method. Subjects were randomly divided into 2 groups. Group A was treated with activity based therapy + baseline therapy and group B was treated with conventional therapy + baseline therapy. 8 subjects in each group. Pre and post treatment evaluation were done by using Spinal cord independence measure scale (SCIM) and International standards for neurological classification of spinal cord injury upper extremity measurement scale (ISNCSCI- UEMS).

Post spinal cord independence measure activity based group mean 26.87±12.87 and conventional group mean 31.50±23.82. The results indicate that conventional therapy and activity based therapy both are helpful in improving upper limb strength and transfer total spinal cord independence measure pre sig.0.96 and post sig.0.57.

Both activity based therapy and conventional therapy equally effective for improving the upper limb strength and transfer in spinal cord injury.

entional therapy.

DETAILED DESCRIPTION:
Spinal cord is the cylindrical structure of nerve fibers and tissues that is enclosed in the spine and provides connection between the brain and all parts of the body. The spinal cord is particularly prone to injury. The spinal cord does not have the ability to repair other parts of the body, if it is damaged. A spinal cord injury happens when the spinal cord is affected by trauma, loss of its normal blood flow, or tumor or infection compression. Lesions in the spinal cord are described as either complete or incomplete.In a complete spinal cord injury, the body suffers complete loss of sensation and muscle control below the injury stage. In an incomplete injury to the spinal cord, there is a certain stay behind feature below injury point. In most cases all sides of the body are similarly affected. Neck injuries to the upper portion of the spinal cord can cause quadriplegia-paralysis of both arms and legs. If the spinal cord injury occurs lower in the back then it can only induce paraplegia-paralysis of both legs. The incidence of SCI to be between 13 and 33 cases per million per year, and their estimate of the incidence of SCI was between 110 and 1120 per million populations. Quadriplegia term refers to the motor and sensory function of cervical spinal cord because neurons inside the neuron damaged the spinal canal. Quadriplegia can cause in the arms, trunk, legs and pelvic organs. Not including brachial plexus or peripheral nervous injury.Trauma is the principal cause of spinal cord injury. Nearly half of the incidents are attributed to accidents involving motor vehicles. Certain forms of trauma include: falling to the spine from a height, stabbing or gunshot wound and sports injuries. Spinal cord damage may also be caused by tumor, infection, or inflammation caused by compression of the spinal cord. Many patients have normal backbone canal and a higher risk of spinal cord injurySome prognostic factors are related to survival, includes demographic, injury, and psychosocial variables. The most important prognostic factors are age and severity of injury including the level of the nervous system, the degree of damage integrity, and ventilator dependence Patients with spinal cord injury (SCI), especially those with higher levels of disease, rely on care and assistance in their daily activities, most of which are provided by informal caregivers. Where home caregivers are involved, low usage of home services is observed. Provides care based on a doctor's prescription based on care needs, assessed by a qualified service provider using standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

* Participants with C6 to T1 tetraplegia.
* Both male and female patients were included
* Participants with traumatic spinal cord injury
* Participants with well oriented behavior were included
* Participants with complete and in complete spinal cord injury
* Participants of all times post injury and any initial sitting were included

Exclusion Criteria:

* Any intervention that measure effectiveness of external devices such as orthotics, frames sittings and chair positions
* Participants with severe neurological disorders, psychological problems and cognitive issues.
* Paraplegic participants or participants involved in gait or walking balance training over ground
* Participants with severe co morbidities and other medical complications
* Participants with pressure ulcers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
SCIM spinal cord independance measure | 6th week
  The Spinal Cord Independence Measure version II (SCIM) was used to assess the ability to accomplish activities of daily living. This scale assesses three areas: (1) self-care (feeding, grooming, bathing, and dressing); (2) respiration and sphincter management; and (3) mobility (bed, transfers, and indoor/outdoor).18 The SCIM III has demonstrated high internal consistency (Cronbach's α = 0.77-0.91) and inter-rater reliability (ICC = 0.96). Moreover, it has shown responsiveness similar to the Functional Independence Measure (FIM).19-21 Ceiling effects were observed in three items: Feeding, Respiration, and Bed mobility, whereas floor effects were observed in 11 items: feeding, bathing (upper and lower body), dressing (upper and lower body), use of toilet, bed mobility, transfers from wheelchair (to bed, toilet, car, and ground), and stair management. changes from the baseline assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Binash afzal, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nas K, Yazmalar L, Sah V, Aydin A, Ones K. Rehabilitation of spinal cord injuries. World J Orthop. 2015 Jan 18;6(1):8-16. doi: 10.5312/wjo.v6.i1.8. eCollection 2015 Jan 18. PMID 25621206
- [Background] Divanoglou A, Trok K, Jorgensen S, Hultling C, Sekakela K, Tasiemski T. Active Rehabilitation for persons with spinal cord injury in Botswana - effects of a community peer-based programme. Spinal Cord. 2019 Oct;57(10):897-905. doi: 10.1038/s41393-019-0300-6. Epub 2019 May 24. PMID 31127198
- [Background] Brogioli M, Schneider S, Popp WL, Albisser U, Brust AK, Velstra IM, Gassert R, Curt A, Starkey ML. Monitoring Upper Limb Recovery after Cervical Spinal Cord Injury: Insights beyond Assessment Scores. Front Neurol. 2016 Aug 31;7:142. doi: 10.3389/fneur.2016.00142. eCollection 2016. PMID 27630612
- [Background] Hachem LD, Ahuja CS, Fehlings MG. Assessment and management of acute spinal cord injury: From point of injury to rehabilitation. J Spinal Cord Med. 2017 Nov;40(6):665-675. doi: 10.1080/10790268.2017.1329076. Epub 2017 Jun 1. PMID 28571527
- [Background] Behrman AL, Ardolino EM, Harkema SJ. Activity-Based Therapy: From Basic Science to Clinical Application for Recovery After Spinal Cord Injury. J Neurol Phys Ther. 2017 Jul;41 Suppl 3(Suppl 3 IV STEP Spec Iss):S39-S45. doi: 10.1097/NPT.0000000000000184. PMID 28628595
- [Background] Quel de Oliveira C, Refshauge K, Middleton J, de Jong L, Davis GM. Effects of Activity-Based Therapy Interventions on Mobility, Independence, and Quality of Life for People with Spinal Cord Injuries: A Systematic Review and Meta-Analysis. J Neurotrauma. 2017 May 1;34(9):1726-1743. doi: 10.1089/neu.2016.4558. Epub 2016 Dec 20. PMID 27809702
- [Background] Argetsinger LC, Singh G, Bickel SG, Calvery ML, Behrman AL. Spinal cord injury in infancy: activity-based therapy impact on health, function, and quality of life in chronic injury. Spinal Cord Ser Cases. 2020 Mar 10;6(1):13. doi: 10.1038/s41394-020-0261-1. PMID 32157078
- [Background] Behrman AL, Argetsinger LC, Roberts MT, Stout D, Thompson J, Ugiliweneza B, Trimble SA. Activity-Based Therapy Targeting Neuromuscular Capacity After Pediatric-Onset Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2019 Spring;25(2):132-149. doi: 10.1310/sci2502-132. PMID 31068745
- [Background] de Oliveira CQ, Middleton JW, Refshauge K, Davis GM. Activity-Based Therapy in a Community Setting for Independence, Mobility, and Sitting Balance for People With Spinal Cord Injuries. J Cent Nerv Syst Dis. 2019 Apr 12;11:1179573519841623. doi: 10.1177/1179573519841623. eCollection 2019. PMID 31019375